CLINICAL TRIAL: NCT07017517
Title: Effect of Physical Therapy on NLRP3 Inflammasome Activation and Muscle Atrophy in Critical Illness Myopathy (PT-NLRP3-CIM).
Brief Title: NLRP3 Inflammasome and Physical Therapy in ICU-Acquired Weakness
Acronym: PT-NLRP3-CIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Collaborators: Clinica Indisa (Other); Hospital de Urgencia y Asistencia Pública (Unknown)
Responsible Party: Principal Investigator, Oscar Arellano, Principal Investigator, PhD Candidate in Biomedical Sciences, University of Chile, University of Chile
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 001-2025
Record Dates: First submitted 2025-05-26; First posted 2025-06-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness Myopathy
Keywords: Critical illness myopathy; Physical therapy; NALP3 inflammasome; Muscle atrophy; ICU-acquired weakness
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced or Additional Physical Therapy Group (Experimental): Critically ill patients at risk of developing CIM will receive enhanced (additional) physical therapy consisting of standard physiotherapy plus servo-assisted lower-limb cycling using the Motomed Letto® device. Therapy will be delivered twice daily, 60 minutes per session, for 7 consecutive days during the early ICU stay. Muscle biopsies from the vastus lateralis will be collected for histological and molecular analyses.
  Interventions: Device: Motomed Letto® servo-assisted cycling + standard physiotherapy
- Conventional Physical Therapy Group (Active Comparator): Critically ill patients at risk of CIM will receive standard physiotherapy delivered according to institutional ICU rehabilitation protocols. The intervention is delivered at the same frequency and clinical stage as the enhanced therapy group.
  Interventions: Behavioral: Standard physiotherapy

INTERVENTIONS:
Device: Motomed Letto® servo-assisted cycling + standard physiotherapy — Servo-assisted cycling using the Motomed Letto® device with a cadence target of 30 revolutions per minute (rpm), performed for 60 minutes twice daily for 7 days. This intervention is administered in addition to standard ICU physiotherapy to critically ill patients at risk of critical illness myopathy (CIM).
  Other Names: Motomed Letto®; Additional Physical Therapy; Enhanced Physical Therapy
  Arms: Enhanced or Additional Physical Therapy Group
Behavioral: Standard physiotherapy — Standard physiotherapy including mobilization and passive/active range-of-motion exercises, delivered during routine ICU care for 7 days.
  Other Names: Conventional physical therapy; routine ICU physiotherapy
  Arms: Conventional Physical Therapy Group

SUMMARY:
The goal of this clinical trial is to study whether physical therapy can reduce NLRP3 inflammasome activation and muscle atrophy in patients with critical illness myopathy (CIM). It will also explore the role of NLRP3 inflammasome in the pathophysiology of CIM.

The main questions this study aims to answer are:

Is NLRP3 inflammasome activation associated with muscle atrophy through the upregulation of atrogenes?

Does physical therapy attenuate NLRP3 inflammasome activation in skeletal muscle, thereby contributing to the prevention or reduction of muscle atrophy in CIM?

Researchers will compare enhanced physical therapy using servo-assisted bed cycling (Motomed Letto®) in critically ill patients at risk of developing CIM during the early phase of ICU stay to conventional physical therapy (standard physiotherapy), to assess whether physical therapy reduces NLRP3 inflammasome activation and muscle degradation.

Participants will:

Be randomized to receive either conventional physical therapy or enhanced physical therapy (Motomed Letto®) for 7 consecutive days. A control group of patients without CIM will also be included.

Undergo assessments of NLRP3 activity, muscle atrophy markers, and transcriptomic profiles from serum and vastus lateralis muscle biopsies.

Be clinically evaluated using the SOFA scale and muscle ultrasound for CIM diagnosis.

Be followed up for changes in muscle strength and physical functionality.

Provide sociodemographic and clinical information to be recorded throughout the study.

DETAILED DESCRIPTION:
Critical illness myopathy (CIM) is a frequent complication in patients admitted to intensive care units (ICUs), characterized by symmetric proximal muscle weakness and respiratory muscle involvement. It has been linked to increased mortality, prolonged hospital stays, and long-term physical disability. CIM may also contribute to post-intensive care syndrome (PICS), which includes persistent cognitive, psychological, and physical impairments. In Chile, approximately 40% of patients with critical illness due to COVID-19 developed this syndrome.

Although several molecular mechanisms have been proposed, the precise etiopathogenesis of CIM remains unclear. Muscle atrophy and contractile dysfunction are hallmark features of CIM. The ubiquitin-proteasome system (UPS) and the upregulation of atrogenes such as MuRF1 and Atrogin-1 have been implicated in its development. In murine models of denervation and sepsis, the NLRP3 inflammasome-a multiprotein complex involved in innate immunity and IL-1β/IL-18 secretion-has been shown to promote muscle atrophy via activation of atrophy-related genes.

Evidence suggests that physical therapy can modulate inflammation at the skeletal muscle level, including downregulation of NLRP3 inflammasome components and IL-1β expression. Mechanical silencing, a major modifiable risk factor in CIM, can be mitigated by early mobilization strategies. However, it remains unknown whether physical therapy directly reduces NLRP3 inflammasome activation and associated muscle atrophy in patients with CIM.

This clinical trial is designed to test the hypothesis that physical therapy decreases NLRP3 inflammasome activity and reduces skeletal muscle atrophy in critically ill patients with CIM. In the early stage of ICU admission, sixteen patients at risk of CIM will be randomized to receive either conventional physical therapy or an enhanced protocol that includes servo-assisted motorized movement therapy (Motomed Letto®), twice daily for 60 minutes. In addition, eight patients without CIM will serve as non-CIM controls.

Muscle biopsy samples from the vastus lateralis will be analyzed to assess histological evidence of muscle atrophy, structural alterations in cellular organelles, and expression of atrophy-related genes. Quantitative real-time PCR (RT-qPCR) will be used to measure mRNA levels of atrogenes, and Western blot will assess protein expression of key mediators of NLRP3 inflammasome signaling. Transcriptomic analysis will be conducted using microarray profiling.

This study will address the following specific aims:

To evaluate the effect of physical therapy on NLRP3 inflammasome activation in skeletal muscle and compare it with non-CIM controls.

To assess the impact of physical therapy on muscle atrophy and explore its relationship with inflammasome activation.

To characterize the gene expression profile of signaling pathways involved in muscle degradation in CIM patients.

To analyze the association between molecular alterations in skeletal muscle and the clinical/ultrasound diagnosis of CIM.

It is expected that enhanced physical therapy will reduce NLRP3 inflammasome activity, attenuate muscle atrophy, and modify gene expression profiles involved in the progression of CIM. These molecular findings are anticipated to correlate with clinical assessments of muscle strength and ultrasound-based diagnosis, supporting the role of early mobilization as a non-pharmacological intervention in the management and prevention of CIM.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of sepsis upon ICU admission.
* Receiving invasive mechanical ventilation with a projected requirement ≥7 days.
* SOFA score ≥8 for three consecutive days within the first five days of ICU admission.

Exclusion Criteria:

* Neurocritical illness.
* Prior malnutrition or cachexia.
* Pre-existing neuromuscular disease.
* Coagulopathy (severe liver disease or continuous dialysis).
* Thrombocytopenia <20,000 platelets/μL.
* Prior Clinical Frailty Scale ≥4.
* Lower limb amputation or fractures.
* Ongoing chemotherapy.
* Pregnancy.
* BMI >35.
* Uncontrolled epilepsy.
* Allergy to ultrasound gel.
* Prior prolonged corticosteroid therapy.
* Expected ICU stay <7 days.
* Imminent death.
* Legal guardian refusal to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Relative mRNA expression of NLRP3, IL-1β, and IL-18 in muscle tissue (RT-qPCR) | Baseline and Day 7 (on the final day of intervention)
  mRNA levels of NLRP3, IL-1β, and IL-18 will be quantified using RT-qPCR from muscle biopsy samples.
Protein expression of phospho-p65S536 and total p65 (Western blot) | Baseline and Day 7 (on the final day of intervention)
  Protein levels of phospho-p65 Serine 536 and total p65 will be assessed by Western blot to evaluate NF-κB pathway activation.
Ratio of cleaved/uncleaved caspase-1, IL-1β, and GSDMD-NT (Western blot) | Baseline and Day 7 (on the final day of intervention)
  Cleaved forms of IL-1β, caspase-1, and GSDMD-NT will be quantified by Western blot and normalized to precursor forms.
Plasma concentrations of IL-1β and IL-18 (ELISA) | Baseline and Day 7 (on the final day of intervention)
  Plasma levels of IL-1β and IL-18 will be measured using ELISA.
Expression of oxidative stress markers and cathepsin B (Western blot) | Baseline and Day 7 (on the final day of intervention)
  Protein carbonylation, nitration, and cathepsin B expression will be analyzed by Western blot.
Expression of cathepsin B (RT-qPCR) | Baseline and Day 7 (on the final day of intervention)
  Cathepsin B expression will be analyzed by RT-qPCR.
Ultrastructural mitochondrial damage and lysosomal vacuolization (TEM) | Baseline and Day 7 (on the final day of intervention)
  Mitochondrial damage and lysosomal vacuole volume will be assessed by transmission electron microscopy.
Muscle fiber diameter (immunofluorescence) | Baseline and Day 7 (on the final day of intervention)
  Fiber diameter in 10 µm cryosections will be measured using anti-laminin immunofluorescence.
mRNA expression of atrogenes: MuRF1, Atrogin-1, MUSA1, TRIM62, TRIM32 | Baseline and Day 7 (on the final day of intervention)
  Atrogene mRNA levels will be quantified using RT-qPCR from muscle biopsies.
Myosin/actin ratio (Western blot) | Baseline and Day 7 (on the final day of intervention)
  Myosin and actin protein levels will be analyzed by Western blot to assess the molecular diagnosis of CIM.
Sarcomeric organization (TEM) | Baseline and Day 7 (on the final day of intervention)
  Evaluation of sarcomeric structure in cryosections using transmission electron microscopy.

SECONDARY OUTCOMES:
Differential expression of genes related to atrophy and inflammasome activation (microarray or nanopore-based RNA sequencing ) | Baseline (prior to intervention) and Day 7 of intervention
  Transcriptomic profiling will be performed using microarray or nanopore-based RNA sequencing to identify changes in gene expression related to CIM and NLRP3 activation.
Correlation between molecular findings and CIM clinical diagnosis | From recovery of consciousness (in ICU or follow-up) through 90-day follow-up
  Correlation analyses will be performed between gene/protein markers and the clinical diagnosis of CIM (based on SOFA score, muscle ultrasound, and clinical assessment with MRC and FSS-ICU scales). Clinical assessments will be conducted once patients regain consciousness, either during ICU stay or follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paola A Llanos, PhD, Study Director — University of Chile
Locations (3):
- Chile (3):
  - Clínica INDISA, Santiago, Metropolitan Region
  - Hospital de Urgencia Asistencia Pública (HUAP), Santiago, Metropolitan Region
  - University of Chile, Santiago, Metropolitan Region

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to uphold ethical standards of patient confidentiality. All data collected will be treated in strict compliance with ethical and regulatory guidelines to protect participant identity. The dissemination of results will occur exclusively in aggregate form, fully anonymized, and only in scientific or academic settings, such as peer-reviewed publications or presentations at conferences.

REFERENCES:
- [Background] Americo-Da-Silva L, Aguilera J, Quinteros-Waltemath O, Sanchez-Aguilera P, Russell J, Cadagan C, Meneses-Valdes R, Sanchez G, Estrada M, Jorquera G, Barrientos G, Llanos P. Activation of the NLRP3 Inflammasome Increases the IL-1beta Level and Decreases GLUT4 Translocation in Skeletal Muscle during Insulin Resistance. Int J Mol Sci. 2021 Sep 23;22(19):10212. doi: 10.3390/ijms221910212. PMID 34638553
- [Background] Neves M Jr, Barreto G, Boobis L, Harris R, Roschel H, Tricoli V, Ugrinowitsch C, Negrao C, Gualano B. Incidence of adverse events associated with percutaneous muscular biopsy among healthy and diseased subjects. Scand J Med Sci Sports. 2012 Apr;22(2):175-8. doi: 10.1111/j.1600-0838.2010.01264.x. Epub 2011 Mar 10. PMID 21392121
- [Background] Raithatha A, Ashraghi MR, Lord C, Limback-Stanic C, Viegas S, Amiras D. Ultrasound-guided muscle biopsy: a practical alternative for investigation of myopathy. Skeletal Radiol. 2020 Nov;49(11):1855-1859. doi: 10.1007/s00256-020-03484-y. Epub 2020 Jun 9. PMID 32519182
- [Background] Kho ME, Molloy AJ, Clarke F, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Pellizzari JR, Tarride JE, Mourtzakis M, Karachi T, Cook DJ; Canadian Critical Care Trials Group. CYCLE pilot: a protocol for a pilot randomised study of early cycle ergometry versus routine physiotherapy in mechanically ventilated patients. BMJ Open. 2016 Apr 8;6(4):e011659. doi: 10.1136/bmjopen-2016-011659. PMID 27059469
- [Background] Moisi L, Mino JC, Guidet B, Vallet H. Frailty assessment in critically ill older adults: a narrative review. Ann Intensive Care. 2024 Jun 18;14(1):93. doi: 10.1186/s13613-024-01315-0. PMID 38888743
- [Background] Mahoney DJ, Carey K, Fu MH, Snow R, Cameron-Smith D, Parise G, Tarnopolsky MA. Real-time RT-PCR analysis of housekeeping genes in human skeletal muscle following acute exercise. Physiol Genomics. 2004 Jul 8;18(2):226-31. doi: 10.1152/physiolgenomics.00067.2004. PMID 15161965
- [Background] Gonzalez-Seguel F, Camus-Molina A, Carcamo M, Hiser S, Needham DM, Leppe J. Inter-observer reliability of trained physiotherapists on the Functional Status Score for the Intensive Care Unit Chilean-Spanish version. Physiother Theory Pract. 2022 Feb;38(2):365-371. doi: 10.1080/09593985.2020.1753272. Epub 2020 Apr 22. PMID 32316800
- [Background] Pardo E, El Behi H, Boizeau P, Verdonk F, Alberti C, Lescot T. Reliability of ultrasound measurements of quadriceps muscle thickness in critically ill patients. BMC Anesthesiol. 2018 Dec 27;18(1):205. doi: 10.1186/s12871-018-0647-9. PMID 30591032
- [Background] Hadda V, Khilnani GC, Kumar R, Dhunguna A, Mittal S, Khan MA, Madan K, Mohan A, Guleria R. Intra- and Inter-observer Reliability of Quadriceps Muscle Thickness Measured with Bedside Ultrasonography by Critical Care Physicians. Indian J Crit Care Med. 2017 Jul;21(7):448-452. doi: 10.4103/ijccm.IJCCM_426_16. PMID 28808365
- [Background] Turan Z, Topaloglu M, Ozyemisci Taskiran O. Medical Research Council-sumscore: a tool for evaluating muscle weakness in patients with post-intensive care syndrome. Crit Care. 2020 Sep 18;24(1):562. doi: 10.1186/s13054-020-03282-x. No abstract available. PMID 32948221
- [Background] Pietrangelo T, Perni S, Di Tano G, Fano-Illic G, Franzini-Armstrong C. A method for the ultrastructural preservation of tiny percutaneous needle biopsy material from skeletal muscle. Int J Mol Med. 2013 Oct;32(4):965-70. doi: 10.3892/ijmm.2013.1454. Epub 2013 Jul 23. PMID 23900509
- [Background] Hodgson CL, Stiller K, Needham DM, Tipping CJ, Harrold M, Baldwin CE, Bradley S, Berney S, Caruana LR, Elliott D, Green M, Haines K, Higgins AM, Kaukonen KM, Leditschke IA, Nickels MR, Paratz J, Patman S, Skinner EH, Young PJ, Zanni JM, Denehy L, Webb SA. Expert consensus and recommendations on safety criteria for active mobilization of mechanically ventilated critically ill adults. Crit Care. 2014 Dec 4;18(6):658. doi: 10.1186/s13054-014-0658-y. PMID 25475522
- [Background] Nickels MR, Aitken LM, Walsham J, Barnett AG, McPhail SM. Critical Care Cycling Study (CYCLIST) trial protocol: a randomised controlled trial of usual care plus additional in-bed cycling sessions versus usual care in the critically ill. BMJ Open. 2017 Oct 22;7(10):e017393. doi: 10.1136/bmjopen-2017-017393. PMID 29061618
- [Background] Kho ME, Berney S, Pastva AM, Kelly L, Reid JC, Burns KEA, Seely AJ, D'Aragon F, Rochwerg B, Ball I, Fox-Robichaud AE, Karachi T, Lamontagne F, Archambault PM, Tsang JL, Duan EH, Muscedere J, Verceles AC, Serri K, English SW, Reeve BK, Mehta S, Rudkowski JC, Heels-Ansdell D, O'Grady HK, Strong G, Obrovac K, Ajami D, Camposilvan L, Tarride JE, Thabane L, Herridge MS, Cook DJ. Early In-Bed Cycle Ergometry in Mechanically Ventilated Patients. NEJM Evid. 2024 Jul;3(7):EVIDoa2400137. doi: 10.1056/EVIDoa2400137. Epub 2024 Jun 12. PMID 38865147
- [Background] Nickels MR, Aitken LM, Barnett AG, Walsham J, King S, Gale NE, Bowen AC, Peel BM, Donaldson SL, Mealing STJ, McPhail SM. Effect of in-bed cycling on acute muscle wasting in critically ill adults: A randomised clinical trial. J Crit Care. 2020 Oct;59:86-93. doi: 10.1016/j.jcrc.2020.05.008. Epub 2020 May 30. PMID 32585438
- [Background] Hough CL, Lieu BK, Caldwell ES. Manual muscle strength testing of critically ill patients: feasibility and interobserver agreement. Crit Care. 2011;15(1):R43. doi: 10.1186/cc10005. Epub 2011 Jan 28. PMID 21276225
- [Background] Wollersheim T, Woehlecke J, Krebs M, Hamati J, Lodka D, Luther-Schroeder A, Langhans C, Haas K, Radtke T, Kleber C, Spies C, Labeit S, Schuelke M, Spuler S, Spranger J, Weber-Carstens S, Fielitz J. Dynamics of myosin degradation in intensive care unit-acquired weakness during severe critical illness. Intensive Care Med. 2014 Apr;40(4):528-38. doi: 10.1007/s00134-014-3224-9. Epub 2014 Feb 15. PMID 24531339
- [Background] Langhans C, Weber-Carstens S, Schmidt F, Hamati J, Kny M, Zhu X, Wollersheim T, Koch S, Krebs M, Schulz H, Lodka D, Saar K, Labeit S, Spies C, Hubner N, Spranger J, Spuler S, Boschmann M, Dittmar G, Butler-Browne G, Mouly V, Fielitz J. Inflammation-induced acute phase response in skeletal muscle and critical illness myopathy. PLoS One. 2014 Mar 20;9(3):e92048. doi: 10.1371/journal.pone.0092048. eCollection 2014. PMID 24651840
- [Background] Mejias-Pena Y, Estebanez B, Rodriguez-Miguelez P, Fernandez-Gonzalo R, Almar M, de Paz JA, Gonzalez-Gallego J, Cuevas MJ. Impact of resistance training on the autophagy-inflammation-apoptosis crosstalk in elderly subjects. Aging (Albany NY). 2017 Feb 2;9(2):408-418. doi: 10.18632/aging.101167. PMID 28160545
- [Background] Ding Y, Xu X. Anti-inflammatory effect of exercise training through reducing inflammasome activation-related inflammatory cytokine levels in overweight/obese populations: A systematic review and meta-analysis. Complement Ther Clin Pract. 2022 Nov;49:101656. doi: 10.1016/j.ctcp.2022.101656. Epub 2022 Aug 28. PMID 36055106
- [Background] Ringleb M, Javelle F, Haunhorst S, Bloch W, Fennen L, Baumgart S, Drube S, Reuken PA, Pletz MW, Wagner H, Gabriel HHW, Puta C. Beyond muscles: Investigating immunoregulatory myokines in acute resistance exercise - A systematic review and meta-analysis. FASEB J. 2024 Apr 15;38(7):e23596. doi: 10.1096/fj.202301619R. PMID 38597350
- [Background] Son WH, Park HT, Jeon BH, Ha MS. Moderate intensity walking exercises reduce the body mass index and vascular inflammatory factors in postmenopausal women with obesity: a randomized controlled trial. Sci Rep. 2023 Nov 17;13(1):20172. doi: 10.1038/s41598-023-47403-2. PMID 37978254
- [Background] Gao K, Su Z, Meng J, Yao Y, Li L, Su Y, Mohammad Rahimi GR. Effect of Exercise Training on Some Anti-Inflammatory Adipokines, High Sensitivity C-Reactive Protein, and Clinical Outcomes in Sedentary Adults With Metabolic Syndrome. Biol Res Nurs. 2024 Jan;26(1):125-138. doi: 10.1177/10998004231195541. Epub 2023 Aug 14. PMID 37579279
- [Background] Wang J, Liu S, Li G, Xiao J. Exercise Regulates the Immune System. Adv Exp Med Biol. 2020;1228:395-408. doi: 10.1007/978-981-15-1792-1_27. PMID 32342473
- [Background] Heidegger CP, Berger MM, Graf S, Zingg W, Darmon P, Costanza MC, Thibault R, Pichard C. Optimisation of energy provision with supplemental parenteral nutrition in critically ill patients: a randomised controlled clinical trial. Lancet. 2013 Feb 2;381(9864):385-93. doi: 10.1016/S0140-6736(12)61351-8. Epub 2012 Dec 3. PMID 23218813
- [Background] Zhang L, Hu W, Cai Z, Liu J, Wu J, Deng Y, Yu K, Chen X, Zhu L, Ma J, Qin Y. Early mobilization of critically ill patients in the intensive care unit: A systematic review and meta-analysis. PLoS One. 2019 Oct 3;14(10):e0223185. doi: 10.1371/journal.pone.0223185. eCollection 2019. PMID 31581205
- [Background] Fuke R, Hifumi T, Kondo Y, Hatakeyama J, Takei T, Yamakawa K, Inoue S, Nishida O. Early rehabilitation to prevent postintensive care syndrome in patients with critical illness: a systematic review and meta-analysis. BMJ Open. 2018 May 5;8(5):e019998. doi: 10.1136/bmjopen-2017-019998. PMID 29730622
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- [Background] Reid JC, Unger J, McCaskell D, Childerhose L, Zorko DJ, Kho ME. Physical rehabilitation interventions in the intensive care unit: a scoping review of 117 studies. J Intensive Care. 2018 Dec 7;6:80. doi: 10.1186/s40560-018-0349-x. eCollection 2018. PMID 30555705
- [Background] Doiron KA, Hoffmann TC, Beller EM. Early intervention (mobilization or active exercise) for critically ill adults in the intensive care unit. Cochrane Database Syst Rev. 2018 Mar 27;3(3):CD010754. doi: 10.1002/14651858.CD010754.pub2. PMID 29582429
- [Background] Chevriaux A, Pilot T, Derangere V, Simonin H, Martine P, Chalmin F, Ghiringhelli F, Rebe C. Cathepsin B Is Required for NLRP3 Inflammasome Activation in Macrophages, Through NLRP3 Interaction. Front Cell Dev Biol. 2020 Mar 31;8:167. doi: 10.3389/fcell.2020.00167. eCollection 2020. PMID 32328491
- [Background] Llano-Diez M, Renaud G, Andersson M, Marrero HG, Cacciani N, Engquist H, Corpeno R, Artemenko K, Bergquist J, Larsson L. Mechanisms underlying ICU muscle wasting and effects of passive mechanical loading. Crit Care. 2012 Oct 26;16(5):R209. doi: 10.1186/cc11841. PMID 23098317
- [Background] Jiroutkova K, Krajcova A, Ziak J, Fric M, Waldauf P, Dzupa V, Gojda J, Nemcova-Furstova V, Kovar J, Elkalaf M, Trnka J, Duska F. Mitochondrial function in skeletal muscle of patients with protracted critical illness and ICU-acquired weakness. Crit Care. 2015 Dec 24;19:448. doi: 10.1186/s13054-015-1160-x. PMID 26699134
- [Background] Vanhorebeek I, Gunst J, Derde S, Derese I, Boussemaere M, Guiza F, Martinet W, Timmermans JP, D'Hoore A, Wouters PJ, Van den Berghe G. Insufficient activation of autophagy allows cellular damage to accumulate in critically ill patients. J Clin Endocrinol Metab. 2011 Apr;96(4):E633-45. doi: 10.1210/jc.2010-2563. Epub 2011 Jan 26. PMID 21270330
- [Background] Cacciani N, Skarlen A, Wen Y, Zhang X, Addinsall AB, Llano-Diez M, Li M, Gransberg L, Hedstrom Y, Bellander BM, Nelson D, Bergquist J, Larsson L. A prospective clinical study on the mechanisms underlying critical illness myopathy-A time-course approach. J Cachexia Sarcopenia Muscle. 2022 Dec;13(6):2669-2682. doi: 10.1002/jcsm.13104. Epub 2022 Oct 12. PMID 36222215
- [Background] Swanson KV, Deng M, Ting JP. The NLRP3 inflammasome: molecular activation and regulation to therapeutics. Nat Rev Immunol. 2019 Aug;19(8):477-489. doi: 10.1038/s41577-019-0165-0. PMID 31036962
- [Background] Liu Y, Wang D, Li T, Yang F, Li Z, Bai X, Wang Y. The role of NLRP3 inflammasome in inflammation-related skeletal muscle atrophy. Front Immunol. 2022 Nov 3;13:1035709. doi: 10.3389/fimmu.2022.1035709. eCollection 2022. PMID 36405697
- [Background] Klaude M, Fredriksson K, Tjader I, Hammarqvist F, Ahlman B, Rooyackers O, Wernerman J. Proteasome proteolytic activity in skeletal muscle is increased in patients with sepsis. Clin Sci (Lond). 2007 Jul;112(9):499-506. doi: 10.1042/CS20060265. PMID 17117920
- [Background] Zanders L, Kny M, Hahn A, Schmidt S, Wundersitz S, Todiras M, Lahmann I, Bandyopadhyay A, Wollersheim T, Kaderali L, Luft FC, Birchmeier C, Weber-Carstens S, Fielitz J. Sepsis induces interleukin 6, gp130/JAK2/STAT3, and muscle wasting. J Cachexia Sarcopenia Muscle. 2022 Feb;13(1):713-727. doi: 10.1002/jcsm.12867. Epub 2021 Nov 24. PMID 34821076
- [Background] Ozdemir M, Bomkamp MP, Hyatt HW, Smuder AJ, Powers SK. Intensive Care Unit Acquired Weakness Is Associated with Rapid Changes to Skeletal Muscle Proteostasis. Cells. 2022 Dec 11;11(24):4005. doi: 10.3390/cells11244005. PMID 36552769
- [Background] Wray CJ, Mammen JM, Hershko DD, Hasselgren PO. Sepsis upregulates the gene expression of multiple ubiquitin ligases in skeletal muscle. Int J Biochem Cell Biol. 2003 May;35(5):698-705. doi: 10.1016/s1357-2725(02)00341-2. PMID 12672461
- [Background] Schmidt F, Kny M, Zhu X, Wollersheim T, Persicke K, Langhans C, Lodka D, Kleber C, Weber-Carstens S, Fielitz J. The E3 ubiquitin ligase TRIM62 and inflammation-induced skeletal muscle atrophy. Crit Care. 2014 Sep 29;18(5):545. doi: 10.1186/s13054-014-0545-6. PMID 25263070
- [Background] Klaude M, Mori M, Tjader I, Gustafsson T, Wernerman J, Rooyackers O. Protein metabolism and gene expression in skeletal muscle of critically ill patients with sepsis. Clin Sci (Lond). 2012 Feb;122(3):133-42. doi: 10.1042/CS20110233. PMID 21880013
- [Background] Constantin D, McCullough J, Mahajan RP, Greenhaff PL. Novel events in the molecular regulation of muscle mass in critically ill patients. J Physiol. 2011 Aug 1;589(Pt 15):3883-95. doi: 10.1113/jphysiol.2011.206193. Epub 2011 Jun 13. PMID 21669975
- [Background] You Z, Huang X, Xiang Y, Dai J, Xu L, Jiang J, Xu J. Ablation of NLRP3 inflammasome attenuates muscle atrophy via inhibiting pyroptosis, proteolysis and apoptosis following denervation. Theranostics. 2023 Jan 1;13(1):374-390. doi: 10.7150/thno.74831. eCollection 2023. PMID 36593964
- [Background] Huang N, Kny M, Riediger F, Busch K, Schmidt S, Luft FC, Slevogt H, Fielitz J. Deletion of Nlrp3 protects from inflammation-induced skeletal muscle atrophy. Intensive Care Med Exp. 2017 Dec;5(1):3. doi: 10.1186/s40635-016-0115-0. Epub 2017 Jan 17. PMID 28097512
- [Background] Walsh CJ, Batt J, Herridge MS, Mathur S, Bader GD, Hu P, Dos Santos CC. Transcriptomic analysis reveals abnormal muscle repair and remodeling in survivors of critical illness with sustained weakness. Sci Rep. 2016 Jul 14;6:29334. doi: 10.1038/srep29334. PMID 27411715
- [Background] Llano-Diez M, Fury W, Okamoto H, Bai Y, Gromada J, Larsson L. RNA-sequencing reveals altered skeletal muscle contraction, E3 ligases, autophagy, apoptosis, and chaperone expression in patients with critical illness myopathy. Skelet Muscle. 2019 Apr 16;9(1):9. doi: 10.1186/s13395-019-0194-1. PMID 30992050
- [Background] Eggelbusch M, Shi A, Broeksma BC, Vazquez-Cruz M, Soares MN, de Wit GMJ, Everts B, Jaspers RT, Wust RCI. The NLRP3 inflammasome contributes to inflammation-induced morphological and metabolic alterations in skeletal muscle. J Cachexia Sarcopenia Muscle. 2022 Dec;13(6):3048-3061. doi: 10.1002/jcsm.13062. Epub 2022 Aug 17. PMID 35978267
- [Background] Antuna E, Potes Y, Baena-Huerta FJ, Cachan-Vega C, Menendez-Coto N, Alvarez Darriba E, Fernandez-Fernandez M, Burgos Bencosme N, Bermudez M, Lopez Alvarez EM, Gutierrez-Rodriguez J, Boga JA, Caballero B, Vega-Naredo I, Coto-Montes A, Garcia-Gonzalez C. NLRP3 Contributes to Sarcopenia Associated to Dependency Recapitulating Inflammatory-Associated Muscle Degeneration. Int J Mol Sci. 2024 Jan 24;25(3):1439. doi: 10.3390/ijms25031439. PMID 38338718
- [Background] Jorquera G, Russell J, Monsalves-Alvarez M, Cruz G, Valladares-Ide D, Basualto-Alarcon C, Barrientos G, Estrada M, Llanos P. NLRP3 Inflammasome: Potential Role in Obesity Related Low-Grade Inflammation and Insulin Resistance in Skeletal Muscle. Int J Mol Sci. 2021 Mar 23;22(6):3254. doi: 10.3390/ijms22063254. PMID 33806797
- [Background] Haberecht-Muller S, Kruger E, Fielitz J. Out of Control: The Role of the Ubiquitin Proteasome System in Skeletal Muscle during Inflammation. Biomolecules. 2021 Sep 8;11(9):1327. doi: 10.3390/biom11091327. PMID 34572540
- [Background] Dos Santos CC, Batt J. ICU-acquired weakness: mechanisms of disability. Curr Opin Crit Care. 2012 Oct;18(5):509-17. doi: 10.1097/MCC.0b013e328357cb5e. PMID 22918258
- [Background] Banduseela VC, Ochala J, Chen YW, Goransson H, Norman H, Radell P, Eriksson LI, Hoffman EP, Larsson L. Gene expression and muscle fiber function in a porcine ICU model. Physiol Genomics. 2009 Nov 6;39(3):141-59. doi: 10.1152/physiolgenomics.00026.2009. Epub 2009 Aug 25. PMID 19706692
- [Background] Banduseela VC, Chen YW, Kultima HG, Norman HS, Aare S, Radell P, Eriksson LI, Hoffman EP, Larsson L. Impaired autophagy, chaperone expression, and protein synthesis in response to critical illness interventions in porcine skeletal muscle. Physiol Genomics. 2013 Jun 17;45(12):477-86. doi: 10.1152/physiolgenomics.00141.2012. Epub 2013 Apr 9. PMID 23572537
- [Background] Gunst J, Derese I, Aertgeerts A, Ververs EJ, Wauters A, Van den Berghe G, Vanhorebeek I. Insufficient autophagy contributes to mitochondrial dysfunction, organ failure, and adverse outcome in an animal model of critical illness. Crit Care Med. 2013 Jan;41(1):182-94. doi: 10.1097/CCM.0b013e3182676657. PMID 23222264
- [Background] Dos Santos C, Hussain SN, Mathur S, Picard M, Herridge M, Correa J, Bain A, Guo Y, Advani A, Advani SL, Tomlinson G, Katzberg H, Streutker CJ, Cameron JI, Schols A, Gosker HR, Batt J; MEND ICU Group; RECOVER Program Investigators; Canadian Critical Care Translational Biology Group. Mechanisms of Chronic Muscle Wasting and Dysfunction after an Intensive Care Unit Stay. A Pilot Study. Am J Respir Crit Care Med. 2016 Oct 1;194(7):821-830. doi: 10.1164/rccm.201512-2344OC. PMID 27058306
- [Background] Batt J, dos Santos CC, Cameron JI, Herridge MS. Intensive care unit-acquired weakness: clinical phenotypes and molecular mechanisms. Am J Respir Crit Care Med. 2013 Feb 1;187(3):238-46. doi: 10.1164/rccm.201205-0954SO. Epub 2012 Nov 29. PMID 23204256
- [Background] Batt J, Herridge MS, Dos Santos CC. From skeletal muscle weakness to functional outcomes following critical illness: a translational biology perspective. Thorax. 2019 Nov;74(11):1091-1098. doi: 10.1136/thoraxjnl-2016-208312. Epub 2019 Aug 20. PMID 31431489
- [Background] Castro-Avila AC, Merino-Osorio C, Gonzalez-Seguel F, Camus-Molina A, Leppe J; IMPACCT COVID-19 study group. Impact on Mental, Physical and Cognitive functioning of a Critical care sTay during the COVID-19 pandemic (IMPACCT COVID-19): protocol for a prospective, multicentre, mixed-methods cohort study. BMJ Open. 2021 Sep 8;11(9):e053610. doi: 10.1136/bmjopen-2021-053610. PMID 34497087
- [Background] Sidiras G, Patsaki I, Karatzanos E, Dakoutrou M, Kouvarakos A, Mitsiou G, Routsi C, Stranjalis G, Nanas S, Gerovasili V. Long term follow-up of quality of life and functional ability in patients with ICU acquired Weakness - A post hoc analysis. J Crit Care. 2019 Oct;53:223-230. doi: 10.1016/j.jcrc.2019.06.022. Epub 2019 Jun 21. PMID 31277049
- [Background] Batt J, Mathur S, Katzberg HD. Mechanism of ICU-acquired weakness: muscle contractility in critical illness. Intensive Care Med. 2017 Apr;43(4):584-586. doi: 10.1007/s00134-017-4730-3. Epub 2017 Mar 3. No abstract available. PMID 28255615
- [Background] Appleton RT, Kinsella J, Quasim T. The incidence of intensive care unit-acquired weakness syndromes: A systematic review. J Intensive Care Soc. 2015 May;16(2):126-136. doi: 10.1177/1751143714563016. Epub 2014 Dec 18. PMID 28979394
- [Background] Weber-Carstens S, Schneider J, Wollersheim T, Assmann A, Bierbrauer J, Marg A, Al Hasani H, Chadt A, Wenzel K, Koch S, Fielitz J, Kleber C, Faust K, Mai K, Spies CD, Luft FC, Boschmann M, Spranger J, Spuler S. Critical illness myopathy and GLUT4: significance of insulin and muscle contraction. Am J Respir Crit Care Med. 2013 Feb 15;187(4):387-96. doi: 10.1164/rccm.201209-1649OC. Epub 2012 Dec 13. PMID 23239154
- [Background] Elkalawy H, Sekhar P, Abosena W. Early detection and assessment of intensive care unit-acquired weakness: a comprehensive review. Acute Crit Care. 2023 Nov;38(4):409-424. doi: 10.4266/acc.2023.00703. Epub 2023 Nov 30. PMID 38052508
- [Background] Hickmann CE, Castanares-Zapatero D, Deldicque L, Van den Bergh P, Caty G, Robert A, Roeseler J, Francaux M, Laterre PF. Impact of Very Early Physical Therapy During Septic Shock on Skeletal Muscle: A Randomized Controlled Trial. Crit Care Med. 2018 Sep;46(9):1436-1443. doi: 10.1097/CCM.0000000000003263. PMID 29957714
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Lad H, Saumur TM, Herridge MS, Dos Santos CC, Mathur S, Batt J, Gilbert PM. Intensive Care Unit-Acquired Weakness: Not just Another Muscle Atrophying Condition. Int J Mol Sci. 2020 Oct 22;21(21):7840. doi: 10.3390/ijms21217840. PMID 33105809
- [Background] Formenti P, Umbrello M, Coppola S, Froio S, Chiumello D. Clinical review: peripheral muscular ultrasound in the ICU. Ann Intensive Care. 2019 May 17;9(1):57. doi: 10.1186/s13613-019-0531-x. PMID 31101987
- [Background] Piva S, Fagoni N, Latronico N. Intensive care unit-acquired weakness: unanswered questions and targets for future research. F1000Res. 2019 Apr 17;8:F1000 Faculty Rev-508. doi: 10.12688/f1000research.17376.1. eCollection 2019. PMID 31069055
- [Background] Friedrich O, Reid MB, Van den Berghe G, Vanhorebeek I, Hermans G, Rich MM, Larsson L. The Sick and the Weak: Neuropathies/Myopathies in the Critically Ill. Physiol Rev. 2015 Jul;95(3):1025-109. doi: 10.1152/physrev.00028.2014. PMID 26133937
- [Background] Bloch S, Polkey MI, Griffiths M, Kemp P. Molecular mechanisms of intensive care unit-acquired weakness. Eur Respir J. 2012 Apr;39(4):1000-11. doi: 10.1183/09031936.00090011. Epub 2011 Sep 29. PMID 21965224
- [Background] Kanova M, Kohout P. Molecular Mechanisms Underlying Intensive Care Unit-Acquired Weakness and Sarcopenia. Int J Mol Sci. 2022 Jul 29;23(15):8396. doi: 10.3390/ijms23158396. PMID 35955530
- [Background] Price DR, Mikkelsen ME, Umscheid CA, Armstrong EJ. Neuromuscular Blocking Agents and Neuromuscular Dysfunction Acquired in Critical Illness: A Systematic Review and Meta-Analysis. Crit Care Med. 2016 Nov;44(11):2070-2078. doi: 10.1097/CCM.0000000000001839. PMID 27513545
- [Background] Latronico N, Herridge M, Hopkins RO, Angus D, Hart N, Hermans G, Iwashyna T, Arabi Y, Citerio G, Ely EW, Hall J, Mehta S, Puntillo K, Van den Hoeven J, Wunsch H, Cook D, Dos Santos C, Rubenfeld G, Vincent JL, Van den Berghe G, Azoulay E, Needham DM. The ICM research agenda on intensive care unit-acquired weakness. Intensive Care Med. 2017 Sep;43(9):1270-1281. doi: 10.1007/s00134-017-4757-5. Epub 2017 Mar 13. PMID 28289812
- [Background] Nakanishi N, Takashima T, Oto J. Muscle atrophy in critically ill patients : a review of its cause, evaluation, and prevention. J Med Invest. 2020;67(1.2):1-10. doi: 10.2152/jmi.67.1. PMID 32378591
- [Background] Schefold JC, Bierbrauer J, Weber-Carstens S. Intensive care unit-acquired weakness (ICUAW) and muscle wasting in critically ill patients with severe sepsis and septic shock. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):147-157. doi: 10.1007/s13539-010-0010-6. Epub 2010 Dec 17. PMID 21475702
- [Background] Yang Z, Wang X, Wang F, Peng Z, Fan Y. A systematic review and meta-analysis of risk factors for intensive care unit acquired weakness. Medicine (Baltimore). 2022 Oct 28;101(43):e31405. doi: 10.1097/MD.0000000000031405. PMID 36316900
- [Background] Tortuyaux R, Davion JB, Jourdain M. Intensive care unit-acquired weakness: Questions the clinician should ask. Rev Neurol (Paris). 2022 Jan-Feb;178(1-2):84-92. doi: 10.1016/j.neurol.2021.12.007. Epub 2022 Jan 5. PMID 34998522
- [Background] Nanas S, Kritikos K, Angelopoulos E, Siafaka A, Tsikriki S, Poriazi M, Kanaloupiti D, Kontogeorgi M, Pratikaki M, Zervakis D, Routsi C, Roussos C. Predisposing factors for critical illness polyneuromyopathy in a multidisciplinary intensive care unit. Acta Neurol Scand. 2008 Sep;118(3):175-81. doi: 10.1111/j.1600-0404.2008.00996.x. Epub 2008 Mar 18. PMID 18355395
- [Background] Rajagopal K, Vijayan D, Thomas SM. Association of SOFA Score with Severity of Muscle Wasting in Critically Ill Patients: A Prospective Observational Study. Indian J Crit Care Med. 2023 Oct;27(10):743-747. doi: 10.5005/jp-journals-10071-24540. PMID 37908434
- [Background] Weber-Carstens S, Deja M, Koch S, Spranger J, Bubser F, Wernecke KD, Spies CD, Spuler S, Keh D. Risk factors in critical illness myopathy during the early course of critical illness: a prospective observational study. Crit Care. 2010;14(3):R119. doi: 10.1186/cc9074. Epub 2010 Jun 18. PMID 20565863
- [Background] Friedrich O, Diermeier S, Larsson L. Weak by the machines: muscle motor protein dysfunction - a side effect of intensive care unit treatment. Acta Physiol (Oxf). 2018 Jan;222(1). doi: 10.1111/apha.12885. Epub 2017 May 3. PMID 28387014
- [Background] Vongchaiudomchoke W, Sathitkarnmanee B, Thanakiattiwibun C, Jarungjitaree S, Chaiwat O. The association between sarcopenia and functional outcomes after hospital discharge among critically ill surgical patients. Asian J Surg. 2022 Jul;45(7):1408-1413. doi: 10.1016/j.asjsur.2021.09.012. Epub 2021 Oct 9. PMID 34635417
- [Background] Rodriguez B, Larsson L, Z'Graggen WJ. Critical Illness Myopathy: Diagnostic Approach and Resulting Therapeutic Implications. Curr Treat Options Neurol. 2022;24(4):173-182. doi: 10.1007/s11940-022-00714-7. Epub 2022 Mar 28. PMID 35370393
- [Background] Mayer KP, Thompson Bastin ML, Montgomery-Yates AA, Pastva AM, Dupont-Versteegden EE, Parry SM, Morris PE. Acute skeletal muscle wasting and dysfunction predict physical disability at hospital discharge in patients with critical illness. Crit Care. 2020 Nov 4;24(1):637. doi: 10.1186/s13054-020-03355-x. PMID 33148301
- [Background] Hrdy O, Vrbica K, Kovar M, Korbicka T, Stepanova R, Gal R. Incidence of muscle wasting in the critically ill: a prospective observational cohort study. Sci Rep. 2023 Jan 13;13(1):742. doi: 10.1038/s41598-023-28071-8. PMID 36639540
- [Background] Giani M, Rezoagli E, Grassi A, Porta M, Riva L, Famularo S, Barbaro A, Bernasconi D, Ippolito D, Bellani G, Braga M, Foti G, Gianotti L, Giani A. Low skeletal muscle index and myosteatosis as predictors of mortality in critically ill surgical patients. Nutrition. 2022 Sep;101:111687. doi: 10.1016/j.nut.2022.111687. Epub 2022 Apr 20. PMID 35700589
- [Background] Yanagi N, Koike T, Kamiya K, Hamazaki N, Nozaki K, Ichikawa T, Matsunaga A, Kuroiwa M, Arai M. Assessment of Sarcopenia in the Intensive Care Unit and 1-Year Mortality in Survivors of Critical Illness. Nutrients. 2021 Aug 8;13(8):2726. doi: 10.3390/nu13082726. PMID 34444886
- [Background] Zhang XM, Chen D, Xie XH, Zhang JE, Zeng Y, Cheng AS. Sarcopenia as a predictor of mortality among the critically ill in an intensive care unit: a systematic review and meta-analysis. BMC Geriatr. 2021 Jun 2;21(1):339. doi: 10.1186/s12877-021-02276-w. PMID 34078275
- [Background] Stibler H, Edstrom L, Ahlbeck K, Remahl S, Ansved T. Electrophoretic determination of the myosin/actin ratio in the diagnosis of critical illness myopathy. Intensive Care Med. 2003 Sep;29(9):1515-27. doi: 10.1007/s00134-003-1894-9. Epub 2003 Aug 12. PMID 12915938
- [Background] Derde S, Hermans G, Derese I, Guiza F, Hedstrom Y, Wouters PJ, Bruyninckx F, D'Hoore A, Larsson L, Van den Berghe G, Vanhorebeek I. Muscle atrophy and preferential loss of myosin in prolonged critically ill patients. Crit Care Med. 2012 Jan;40(1):79-89. doi: 10.1097/CCM.0b013e31822d7c18. PMID 21926599
- [Background] Wilcox SR. Corticosteroids and neuromuscular blockers in development of critical illness neuromuscular abnormalities: A historical review. J Crit Care. 2017 Feb;37:149-155. doi: 10.1016/j.jcrc.2016.09.018. Epub 2016 Sep 26. PMID 27736708
- [Background] Stevens RD, Marshall SA, Cornblath DR, Hoke A, Needham DM, de Jonghe B, Ali NA, Sharshar T. A framework for diagnosing and classifying intensive care unit-acquired weakness. Crit Care Med. 2009 Oct;37(10 Suppl):S299-308. doi: 10.1097/CCM.0b013e3181b6ef67. PMID 20046114
- [Background] Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, Hopkins RO, Hough CL, Kress JP, Latronico N, Moss M, Needham DM, Rich MM, Stevens RD, Wilson KC, Winkelman C, Zochodne DW, Ali NA; ATS Committee on ICU-acquired Weakness in Adults; American Thoracic Society. An official American Thoracic Society Clinical Practice guideline: the diagnosis of intensive care unit-acquired weakness in adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437-46. doi: 10.1164/rccm.201411-2011ST. PMID 25496103
- [Background] Barreiro E. Models of disuse muscle atrophy: therapeutic implications in critically ill patients. Ann Transl Med. 2018 Jan;6(2):29. doi: 10.21037/atm.2017.12.12. PMID 29430446
- [Background] Wang W, Xu C, Ma X, Zhang X, Xie P. Intensive Care Unit-Acquired Weakness: A Review of Recent Progress With a Look Toward the Future. Front Med (Lausanne). 2020 Nov 23;7:559789. doi: 10.3389/fmed.2020.559789. eCollection 2020. PMID 33330523
- [Background] Schefold JC, Wollersheim T, Grunow JJ, Luedi MM, Z'Graggen WJ, Weber-Carstens S. Muscular weakness and muscle wasting in the critically ill. J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1399-1412. doi: 10.1002/jcsm.12620. Epub 2020 Sep 7. PMID 32893974
- [Background] Kress JP, Hall JB. ICU-acquired weakness and recovery from critical illness. N Engl J Med. 2014 Apr 24;370(17):1626-35. doi: 10.1056/NEJMra1209390. No abstract available. PMID 24758618
- [Background] Chen J, Huang M. Intensive care unit-acquired weakness: Recent insights. J Intensive Med. 2023 Aug 30;4(1):73-80. doi: 10.1016/j.jointm.2023.07.002. eCollection 2024 Jan. PMID 38263973
- [Background] Vanhorebeek I, Latronico N, Van den Berghe G. ICU-acquired weakness. Intensive Care Med. 2020 Apr;46(4):637-653. doi: 10.1007/s00134-020-05944-4. Epub 2020 Feb 19. PMID 32076765
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Z'Graggen WJ, Tankisi H. Critical Illness Myopathy. J Clin Neurophysiol. 2020 May;37(3):200-204. doi: 10.1097/WNP.0000000000000652. PMID 32358245

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT07017517/Prot_SAP_002.pdf
  • Informed Consent Form: All IFC (2025-08-11): https://cdn.clinicaltrials.gov/large-docs/17/NCT07017517/ICF_003.pdf